CLINICAL TRIAL: NCT01987765
Title: Safety and Efficacy of Relestat Ophthalmic Solution 0.05% for Allergic Conjunctivitis in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 198027-A
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relestat Ophthalmic Solution 0.05%: Patients who are prescribed Relestat Ophthalmic Solution 0.05% as local standard of care in clinical practice.
  Interventions: Drug: Relestat Ophthalmic Solution 0.05%

INTERVENTIONS:
Drug: Relestat Ophthalmic Solution 0.05% — Relestat Ophthalmic Solution 0.05% prescribed as local standard of care in clinical practice.

SUMMARY:
This study is a Post-Marketing Surveillance study in Korea to evaluate the safety and efficacy of Relestat Ophthalmic Solution 0.05% in patients with allergic conjunctivitis who are treated with Relestat as standard of care in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Allergic Conjunctivitis treated with Relestat Ophthalmic Solution in clinical practice.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Allergic Conjunctivitis treated with Relestat Ophthalmic Solution in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Gangwon-do, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Relestat Ophthalmic Solution 0.05%
Started | 847
Completed | 745
Not Completed | 102
Not completed — Protocol Violation | 65
Not completed — Lost to Follow-up | 37

BASELINE CHARACTERISTICS:
Population: The Safety Assessment Population which included all patients who completed the study, was used for the analysis of baseline characteristics.
Arm/Group | Relestat Ophthalmic Solution 0.05%
Number analyzed (Participants) | 745
Age, Customized [Number; unit: Participants]
  <20 years | 143
  20 to 29 years | 129
  30 to 39 years | 139
  40 to 49 years | 127
  50 to 59 years | 84
  60 to 69 years | 73
  ≥70 years | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 487
  Male | 258

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Reporting Adverse Events
Description: An adverse event is any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: Up to 10 Months
Population: Safety Assessment Population: included all patients who completed the study.
Measure: Number; unit: Percentage of Patients
Arm/Group | Relestat Ophthalmic Solution 0.05%
Number analyzed (Participants) | 745
Percentage of Patients | 0.13

2. Primary Outcome: Change From Baseline in Eye Symptoms Total Score on a 4-Point Scale
Description: Itchiness, conjunctival hyperaemia (redness), lacrimation (tearing), and foreign body sensation were each evaluated on a 4-point scale ranging from 0 (best) to 3 (worst). The eye symptom total score is the sum of the individual symptom scores and ranges from 0 (best) to 12 (worst). A negative number change from baseline indicates an improvement.
Time Frame: Baseline, 2 Weeks
Population: Efficacy Assessment Population: included all patients in the Safety Assessment Population whose data was available for analysis.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Relestat Ophthalmic Solution 0.05%
Number analyzed (Participants) | 741
Scores on a Scale
  Baseline | 5.58 (2.25)
  Change from Baseline at 2 Weeks | -4.06 (2.17)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during follow-up, for a period of up to 10 months.
Description: The Safety Assessment Population was used to assess adverse events (AEs) and serious adverse events (SAE). The Safety Assessment Population included all patients who completed the study.
Arm/Group | Relestat Ophthalmic Solution 0.05%
Serious Adverse Events (participants affected / at risk) | 0/745
Other Adverse Events (participants affected / at risk) | 0/745

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.